CLINICAL TRIAL: NCT00926848
Title: Reducing Risk in Cardiac Rehabilitation: Partners Together in Health (PaTH) Intervention Study
Acronym: PaTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0544-08-FB; 1R15NR010923-01A1 (NIH)
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Coronary Heart Disease; Cardiac Rehabilitation
Keywords: coronary heart disease; cardiac rehabilitation; lifestyle change; coronary artery bypass graft; social support; social cognitive learning theory
MeSH Terms: conditions — Coronary Disease | interventions — Health; Methods

STUDY DESIGN:
Intervention Model Description: Patients and partners in the PaTH intervention group formally joined and participated in the full cardiac rehabilitation (CR) program consisting of 18-36 exercise and 18 educational sessions. In the usual care group, only patients received the exercise and educational sessions; partners received the educational sessions only.
Who Masked: Outcomes Assessor
Masking Description: The research personnel who were collecting outcomes data were unaware of the subjects' group assignment.
Oversight: Data Monitoring Committee: No

ARMS (2):
- PaTH intervention group (Experimental): The PaTH intervention group for patients and partners consisted of participation in a structured and formal cardiac rehabilitation program:
  * 18-36 exercise sessions
  * 18 educational sessions. The intervention consisted of patients and partners participating together in a formal cardiac rehabilitation program when typically just patients participate. In addition, partners were asked to make the same healthy eating and exercise changes that patients did to meet guidelines for health.
  Interventions: Behavioral: Partners Together in Health (PaTH) Intervention
- Usual care group (Active Comparator): The usual care group intervention for patients only consisted of participation in a structured and formal cardiac rehabilitation program:
  * 18-36 exercise sessions and 18 educational sessions
  Partners participated in the 18 educational sessions only.
  Interventions: Behavioral: Partners Together in Health (PaTH) Intervention

INTERVENTIONS:
Behavioral: Partners Together in Health (PaTH) Intervention — Patients and partners in the PaTH experimental group participated in 18-36 exercise and 18 educational sessions in a structured cardiac rehabilitation program. Patients in the Usual care group also participated in 18-36 exercise and 18 educational sessions; partners, however, only participated in the educational sessions.

SUMMARY:
The objective of the proposed study, using an experimental, two-group (n = 30 couples in each group) repeated measures design, was to pilot test the effects of the PaTH Intervention versus a usual care group in improving the following outcomes: a) physical activity and healthy eating behaviors, and b) functional capacity. The primary outcomes will be physical activity behavior (minutes per week) and eating behavior (percent saturated fat) at the 6 month time point in both the coronary artery bypass graft (CABG) patient and his/her partner. Secondary outcome includes functional capacity in patients and partners at 6 months.

DETAILED DESCRIPTION:
Long-term maintenance of lifestyle changes to reduce cardiovascular risk factors after coronary artery bypass graft (CABG) surgery is essential to positively influence health outcomes. Despite proven efficacy of cardiac rehabilitation (CR) in helping patients initiate lifestyle changes, less than 50% of CABG patients maintain lifestyle changes by 6 months post-CABG. It is known that the spouse is the main source of social support for the recovering cardiac patient and frequently attends cardiac rehabilitation with the patient to provide transportation, emotional support, or attend educational classes. In spite of these supportive behaviors, however; adherence still drops off after CR. Lifestyle interventions that specifically target the marital partners as a unit may be more efficacious than current individually-oriented education strategies. The objective of the proposed feasibility study, using an experimental, two-group (n = 30 couples in each group) repeated measures design, will be to pilot test the effects of the Partners Together in Health (PaTH) Intervention versus usual care in improving physical activity and healthy eating behaviors, and functional capacity. The specific aims are to assess the feasibility of implementing the PaTH Intervention and generate pilot data on all outcome variables in both the CABG patient and the partner to estimate effect sizes needed to determine the sample size requirements for the larger study. Partners in the PaTH Intervention group will formally join CR with the patient to participate in exercise sessions and educational classes to undertake comprehensive risk reduction for themselves, and to make the same positive physical activity/exercise and healthy eating lifestyle changes as the patient. Partners in the usual care group will be invited to attend the educational sessions with the patient as is currently usual care. The primary outcomes will be physical activity behavior (minutes per week) and eating behavior (percent saturated fat) at the 6 month time point in both the coronary artery bypass graft (CABG) patient and his/her partner. The secondary outcome includes functional capacity in patients and partners at 6 months. The PaTH intervention is innovative because it allows the couple to build new habits together so they can motivate and support one another on their journey toward health, it uses an existing, well-established treatment method (cardiac rehab) to deliver cost-effective care (Balady et al., 2007), it provides self-efficacy and social support for both members of the dyad in making behavioral changes, and no other studies testing the effects of including the partner in CR were found.

ELIGIBILITY:
Inclusion Criteria:

* age 19 or older
* diagnosis of first-time coronary artery bypass graft surgery (CABGs) and enrollment in outpatient CR
* married or living with partner for more than 1 year
* partner is also willing to participate
* no history of psychiatric illness
* classified as low to moderate risk for the occurrence of cardiac events during exercise (AACVPR, 2004).
* first-time CABG patients

Eligible partners will:

* be age 19 or older
* have no history of psychiatric illness
* be classified as low to moderate risk for the occurrence of cardiac events during exercise
* have written permission from the partner's primary health care provider to participate in the study.

Exclusion Criteria:

* orthopedic problems that would prevent them from walking or exercising
* history of cardiac arrest, sudden death, complex dysrhythmias at rest, or CHF diagnosis
* resting systolic BP > 200 mmHg or diastolic BP > 100 mmHg
* a concomitant diagnosis or procedure such as valve repair/replacement or aneurysmectomy
* debilitating non-cardiac disease such as renal failure or anemia
* severe chronic obstructive lung disease (FEV1 < 1 liter)
* poorly controlled diabetics (diagnosed with diabetic ketoacidosis within the past 6 months or a current HgA1c > 11).

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2012-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernice C Yates, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 158 couples were assessed for eligibility; 87 couples did not meet inclusion criteria. Of the 72 eligible, 37 declined to participate. Of the 34 couples who consented, 17 couples (17 patients and 17 partners) were randomly allocated to the PaTH group and 17 couples (17 patients and 17 partners) to the usual care group = 68 individual participants.
Pre-assignment Details: One patient in the PaTH intervention group did not tolerate the baseline (T1) exercise treadmill test due to orthopedic problems. Thus, this couple was ineligible to continue in the study.
Groups:
- Usual Care Group: In the usual care group, only patients received the full cardiac rehabilitation program consisting of comprehensive risk reduction, educational classes, and 3 exercise sessions per week for 8 weeks. Partners participated in the educational classes only.
- PaTH Intervention Group: Patients and partners in the PaTH intervention group formally joined and participated in the full cardiac rehabilitation (CR) program consisting of comprehensive risk reduction educational classes and 3 exercise sessions/week for 8 weeks. These CR components were: prescribed exercise, education about cardiac risk factor modification, and counseling about self-efficacy strategies that may be effective in assisting with initial lifestyle changes and in preventing and managing relapse. All patients and partners in CR will be provided with a comprehensive, individualized, multidisciplinary risk factor modification program focused on all of the person's risk factors for coronary heart disease.
Period: Overall Study
Arm/Group | Usual Care Group | PaTH Intervention Group
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PaTH Intervention Group: Patients and partners participated in 18-36 exercise and 18 educational sessions.
- Usual Care Group: Only patients participated in 18-36 exercise and 18 educational sessions. Partners only participated in educational sessions.
- Total: Total of all reporting groups
Arm/Group | PaTH Intervention Group | Usual Care Group | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10.3) | 59.5 (14.1) | 60.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 17 | 16 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 32 | 32 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 34 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Healthy Lifestyle Behavior Was Physical Activity/Exercise in Patients
Description: Physical activity/exercise behavior was measured using an Actigraph accelerometer at 6 months.
Time Frame: 6 months post enrollment/baseline
Measure: Mean (Standard Deviation); unit: minutes per day
Groups:
- PaTH Intervention Group (Patients Only, n=17): Patients in the PaTH intervention group formally joined and participated in the full cardiac rehabilitation (CR) program consisting of comprehensive risk reduction educational classes and 3 exercise sessions/week for 8 weeks.
- Usual Care Group (Patients Only, n=17): In the usual care group, only patients received the full cardiac rehabilitation program consisting of comprehensive risk reduction, educational classes, and 3 exercise sessions per week for 8 weeks. Partners participated in the educational classes only.
Arm/Group | PaTH Intervention Group (Patients Only, n=17) | Usual Care Group (Patients Only, n=17)
Number analyzed (Participants) | 17 | 17
minutes per day | 25.8 (3.3) | 21.8 (3.4)
Statistical Analysis 1: Comparison: PaTH Intervention Group (Patients Only, n=17) vs Usual Care Group (Patients Only, n=17); Test type: Superiority; p > .05, t-test, 2 sided; Mean Difference (Final Values) = 4.0

2. Primary Outcome: Healthy Lifestyle Behavior Was Physical Activity/Exercise in Partners
Description: Physical activity/exercise behavior was measured using an Actigraph accelerometer at 6 months.
Time Frame: 6 months post enrollment/baseline
Measure: Mean (Standard Deviation); unit: minutes per day
Groups:
- PaTH Intervention Group (Partners Only, n=17): Partners in the PaTH intervention group participated in 18-36 exercise sessions and 18 educational sessions.
- Usual Care Group (Partners Only, n=17): In the usual care group, partners participated in 18 educational sessions.
Arm/Group | PaTH Intervention Group (Partners Only, n=17) | Usual Care Group (Partners Only, n=17)
Number analyzed (Participants) | 17 | 17
minutes per day | 45.0 (4.6) | 38.4 (5.8)
Statistical Analysis 1: Comparison: PaTH Intervention Group (Partners Only, n=17) vs Usual Care Group (Partners Only, n=17); Test type: Superiority; p > .05, t-test, 2 sided; Mean Difference (Final Values) = 6.6

3. Primary Outcome: Eating Behavior (% Saturated Fat) in Patients
Description: Eating behavior (% saturated fat) was measured using a 3-day food record.
Time Frame: 6 months post baseline
Measure: Mean (Standard Deviation); unit: percent saturated fat per day
Groups:
- PaTH Intervention Group (Patients Only): Patients in the PaTH intervention group participated in 18-36 exercise sessions and 18 educational sessions.
- Usual Care Group (Patients Only): The usual care group intervention for patients only consisted of participation in 18-36 exercise sessions and 18 educational sessions. Partners participated in the 18 educational sessions only.
Arm/Group | PaTH Intervention Group (Patients Only) | Usual Care Group (Patients Only)
Number analyzed (Participants) | 17 | 17
percent saturated fat per day | 10.0 (2.4) | 10.3 (2.6)
Statistical Analysis 1: Comparison: PaTH Intervention Group (Patients Only) vs Usual Care Group (Patients Only); Test type: Superiority; p > .05, t-test, 2 sided; Mean Difference (Final Values) = 0.3

4. Primary Outcome: Eating Behavior (% Saturated Fat) in Partners
Description: Eating behavior (% saturated fat) was measured using a 3-day food record.
Time Frame: 6 months post baseline
Measure: Mean (Standard Deviation); unit: percent saturated fat per day
Groups:
- PaTH Intervention Group (Partners Only): Partners in the PaTH intervention group participated in 18-36 exercise sessions and 18 educational sessions.
- Usual Care Group (Partners Only): Partners in the usual care group participated in the 18 educational sessions only.
Arm/Group | PaTH Intervention Group (Partners Only) | Usual Care Group (Partners Only)
Number analyzed (Participants) | 17 | 17
percent saturated fat per day | 10.6 (2.3) | 11.2 (2.3)
Statistical Analysis 1: Comparison: PaTH Intervention Group (Partners Only) vs Usual Care Group (Partners Only); Test type: Superiority; p > .05, t-test, 2 sided; Mean Difference (Final Values) = 0.6

5. Secondary Outcome: Functional Capacity in Patients
Description: Exercise tolerance test using a treadmill
Time Frame: 6 months post baseline
Measure: Mean (Standard Deviation); unit: Metabolic equivalents (METs)
Groups:
- PaTH Intervention Group (Patients Only): The PaTH intervention group for patients and partners consisted of participation in a structured and formal cardiac rehabilitation program:
  * 18-36 exercise sessions
  * 18 educational sessions
- Usual Care Group (Patients Only): The usual care group intervention for patients only consisted of participation in a structured and formal cardiac rehabilitation program:
  * 18-36 exercise sessions and 18 educational sessions
  Partners participated in the 18 educational sessions only.
Arm/Group | PaTH Intervention Group (Patients Only) | Usual Care Group (Patients Only)
Number analyzed (Participants) | 17 | 17
Metabolic equivalents (METs) | 9.8 (1.7) | 9.5 (1.9)
Statistical Analysis 1: Comparison: PaTH Intervention Group (Patients Only) vs Usual Care Group (Patients Only); Test type: Superiority; p > .05, t-test, 2 sided; Mean Difference (Final Values) = 0.3

6. Secondary Outcome: Functional Capacity in Partners
Description: Exercise tolerance test using a treadmill
Time Frame: 6 months post baseline
Measure: Mean (Standard Deviation); unit: Metabolic equivalents (METs)
Groups:
- PaTH Intervention Group (Partners): The PaTH intervention group for patients and partners consisted of participation in a structured and formal cardiac rehabilitation program:
  * 18-36 exercise sessions
  * 18 educational sessions
- Usual Care Group (Partners): The usual care group intervention for patients only consisted of participation in a structured and formal cardiac rehabilitation program:
  * 18-36 exercise sessions and 18 educational sessions
  Partners participated in the 18 educational sessions only.
Arm/Group | PaTH Intervention Group (Partners) | Usual Care Group (Partners)
Number analyzed (Participants) | 17 | 17
Metabolic equivalents (METs) | 10.3 (1.8) | 9.5 (2.0)
Statistical Analysis 1: Comparison: PaTH Intervention Group (Partners) vs Usual Care Group (Partners); Test type: Superiority; p > .05, t-test, 2 sided; Mean Difference (Final Values) = 0.8

ADVERSE EVENTS:
Groups:
- PaTH Intervention Group: Patients and partners in the PaTH intervention group formally joined and participated in the full cardiac rehabilitation (CR) program consisting of comprehensive risk reduction educational classes and 3 exercise sessions/week for 8 weeks.
Arm/Group | PaTH Intervention Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 1/32 | 0/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PaTH Intervention Group (N=32) | Usual Care Group (N=32)
orthopedic pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 — Hip pain 3 days post exercise test

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No